CLINICAL TRIAL: NCT00745446
Title: The Effect of a Retrofit Particle Trap on the Vascular Effects of Diesel Exhaust Inhalation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Umeå University (Other)
Responsible Party: Dr Anders Blomberg, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VOLVO 3ARM
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Heart Disease
Keywords: Air pollution; Diesel exhaust; Endothelial function; Vascular function; Particle trap; Thrombosis; effects; inhalation
MeSH Terms: conditions — Heart Diseases; Thrombosis; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 1 hour exposure to filtered air
  Interventions: Procedure: Forearm Venous Occlusion Plethysmography
- 2 (Experimental): 1 hour exposure to diesel exhaust (300mcg/m3)
  Interventions: Procedure: Forearm Venous Occlusion Plethysmography
- 3 (Experimental): 1 hour exposure to filtered diesel exhaust
  Interventions: Procedure: Forearm Venous Occlusion Plethysmography

INTERVENTIONS:
Procedure: Forearm Venous Occlusion Plethysmography — Forearm venous occlusion plethysmography with intra-arterial infusion of Acetylcholine (5-20mcg/min), bradykinin (30-300mcg/min), sodium nitroprusside (2-8mcg/min) and Verapamil (2-10 mcg/min) into non-dominant brachial artery

SUMMARY:
The purpose of this study is to determine whether a retrofit particle trap can reduce the adverse vascular responses to diesel exhaust inhalation

DETAILED DESCRIPTION:
18 subjects healthy male volunteers will be recruited at Umeå University. In a randomised, double blind 3 way crossover trial, subjects will be exposed to filtered air, diesel exhaust (300mcg/m3) or filtered diesel exhaust for 1 hour during intermittent exercise.

2 hours following the exposure, thrombogenicity will be assessed using the Badimon chamber - an ex-vivo model of thrombosis formed under constant flow conditions.

Forearm blood flow in response to infused intra-brachial vasodilators will be measured using venous occlusion plethysmography 6 hours after the exposure.

Arterial stiffness will be measured using peripheral arterial applanation tonometry in the hour post-exposure.

Blood samples will be collected at timepoints over the 24 hours after exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Intercurrent illness
* Smoking
* Significant occupational exposure to air pollution
* Regular medication usage

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow in response to infused intra-arterial vasodilators | 6 hours post-exposure

SECONDARY OUTCOMES:
Arterial stiffness measured by applanation tonometry | In the 1 hour following exposure
Thrombogenicity measured using the Badimon chamber - an ex-vivo model of thrombosis under conditions of continuous flow | 2 hours after the exposure
Exhaled nitric oxide - a marker of pulmonary inflammation | 1 hour & 6 hours after exposure
Endogenous fibrinolytic capacity - measured as net release of t-PA in response to infused bradykinin | 6 hours after exposure
Biochemical markers of systemic inflammation | Baseline, 2, 6 & 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anders Blomberg, MD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Västerbottens, Sweden

REFERENCES:
- [Derived] Lucking AJ, Lundback M, Barath SL, Mills NL, Sidhu MK, Langrish JP, Boon NA, Pourazar J, Badimon JJ, Gerlofs-Nijland ME, Cassee FR, Boman C, Donaldson K, Sandstrom T, Newby DE, Blomberg A. Particle traps prevent adverse vascular and prothrombotic effects of diesel engine exhaust inhalation in men. Circulation. 2011 Apr 26;123(16):1721-8. doi: 10.1161/CIRCULATIONAHA.110.987263. Epub 2011 Apr 11. PMID 21482966